CLINICAL TRIAL: NCT02308306
Title: Predictive Markers of the Effects of Opioid Therapy in Opioid naïve Patients With Chronic Pain: an International, Multi-centre, Observational Cohort Study (ABILITY)
Brief Title: Predictive Markers of the Effects of Opioid Therapy
Acronym: ABILITY
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: ABILITY
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Opioid Analgesic Treatment Response; Chronic Pain
Keywords: Chronic pain; Opioid analgesics; Prediction study; Pharmaco-EEG
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Opioid analgesics: Opioid treatment is determined, prescribed, modified and discontinued at the sole discretion of the treating physician at each research site; regardless of generic name, manufacturer, constituent components, route of administration, and dosing schedule (including titration and run-in periods).

SUMMARY:
The overall goal of the ABILITY study is to help improve pain diagnostics and treatment by developing an implementable clinical computerised decision support system based on individual patient characteristics.

The investigators hypothesize that successful pain control with opioids can be predicted before treatment initiation with advanced data analyses of data originating from pre-treatment EEG, QST and pain-related catastrophic thinking.

The primary objective of this study is the identification of markers that can be used to individualize treatment recommendations, i.e. to reliably predict the response of pain to opioids.

Markers are selected among the most promising data and machine-learning methods are used for the prediction. This includes determining the associations between a battery of selected pre-treatment clinical predictive markers and the analgesic effect of opioid treatment in opioid naïve chronic pain patients, including indication and responder identification.

The key secondary objectives are as follows: to investigate pre-treatment clinical predictive markers as predictors of opioid treatment efficacy and effectiveness in terms of the following:

* Pain intensity and unpleasantness
* Use of rescue analgesics
* Physical functioning
* Global improvement and satisfaction with treatment

ELIGIBILITY:
Inclusion Criteria:

* Pain duration ≥ 3 months.
* Minimum baseline pain intensity ≥ 4 on a 0-10 numerical rating scale (over the past week).
* Maximum baseline pain intensity < 9 on a 0-10 numerical rating scale (over the past week).
* Prescribed opioid treatment (ATC: N02)
* Anticipated to stay on prescribed opioid treatment throughout the study, i.e. >14 days.
* Anticipated to stay on any concomitant non-opioid treatment throughout the study, i.e. >14 days.
* Subject may be male or female, age >18 years old.
* Is willing and able to comply with study procedures as judged by the site investigator.
* Subject has voluntarily signed and dated the study-specific informed consent form, approved by an Independent Ethics Committee, after the nature of the study has been explained and the subject has had the opportunity to ask questions. The informed consent form must be signed before any study-specific procedures are performed.

Exclusion Criteria:

* Has a mental incapacity or language barriers precluding adequate understanding of study procedures.
* Is considered by the site investigator unsuitable to participate in the study for any other reason, for instance due to a significant serious underlying condition.
* Recently received opioids on a daily basis (within the last 10 weeks).
* Current alcohol or substance abuse, according to the site investigator's medical judgement.
* Is anticipated to undergo a painful procedure(s) (e.g. surgery) during the study, which can interfere with the experience of the chronic pain condition for which the subject is to receive opioids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with an insufficiently treated chronic pain condition (with non-opioids ± adjuvants), and expected to benefit from the administration of opioids (as necessary) to obtain freedom from pain.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Reduction of chronic pain assessed by 0-10 numerical rating scale (NRS) scores | After 14-days of opioid treatment
  The absolute and percentage change from baseline in ratings of average pain in the past week at Day 14. Of note, a percentage change of ≥30% is considered clinically significant.
Improvement of health-related quality of life assessed by QLQ-C30 scores | After 14 days of opioid treatment
  The absolute and percentage change from baseline in ratings of health-related quality of life in the past week at Day 14. A subjectively significant change in QLQ-C30 scores is one that is ≥10 from baseline.

SECONDARY OUTCOMES:
BPI worst pain in the past week | Day 14 post-treatment
  Change from baseline
BPI least pain in the past week | Day 14 post-treatment
  Change from baseline
BPI current pain in the past week | Day 14 post-treatment
  Change from baseline
BPI pain severity in the past week | Day 14 post-treatment
  Change from baseline
BPI pain interference score | Day 14 post-treatment
  Change from baseline
Improvement score | Day 14 post-treatment
  Proportion with score >4
Concomitant and rescue medication | Until 14 days post-treatment
Adverse events | Until 14 days post-treatment
  Number (%) of the following:
  1. Constipation
  2. Dry mouth
  3. Nausea/Vomiting
  4. Sedation
  5. Sweats
  6. Bad dreams
  7. Dysphoria/Delirium
  8. Myoclonus/Seizures
  9. Pruritus/Urticaria
  10. Urinary retention

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn M Drewes, MD, PhD, DMSci, Study Chair — Aalborg University Hospital, Denmark; Anne E Olesen, MSc (Pharm), PhD, Study Director — Aalborg University Hospital, Denmark; Kasper Grosen, MHSc, PhD, Study Director — Aarhus University / Aarhus University Hospital, Denmark; Mogens Pfeiffer-Jensen, MD, PhD, Principal Investigator — Aarhus University Hospital, Denmark; Michael Kamp-Jensen, MD, PhD, Principal Investigator — Hospitalet Valdemar, Denmark; Bart Morlion, MD, PhD, Principal Investigator — University of Leuven / University Hospitals Leuven, Belgium; Gorazd Pozlep, MD, Principal Investigator — Ljubljana University Medical Centre, Slovenia; Torsten Jonsson, MD, Principal Investigator — Hospitalet Valdemar, Denmark
Locations (5):
- KU Leuven and the Leuven Centre for Algology & Pain Management, Leuven, Pellenberg, Belgium
- Denmark (3):
  - Friklinikken, Give, Give
  - Department of Rheumatology, Aarhus University Hospital, Aarhus C
  - Hospitalet Valdemar, Ringsted
- Ljubljana University Medical Centre, Department of Anaesthetics and Surgical Intensive Care, Ljubljana, Slovenia

REFERENCES:
- See also: Related Info — http://www.mech-sense.com